CLINICAL TRIAL: NCT01343095
Title: A Randomized Controlled Trial of Direct Noise Reduction in the ICU Using Overnight Application of In-ear Earplugs or In-ear Earplugs Plus Noise-Canceling Headphones to Reduce the Incidence and Duration of ICU Delirium
Brief Title: Direct Noise Reduction in the Intensive Care Units (ICU) Using Earplugs and Noise Canceling Headphones
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Loss of study staff
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00013140
Record Dates: First submitted 2011-04-13; First posted 2011-04-27 (Estimated); Results first posted 2017-12-20 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-08

CONDITIONS: Delirium; Sleep Fragmentation
Keywords: ICU Delirium; Delirium; Sleep Quality; Sleep Efficiency; ICU Noise; Noise Reduction; Earplugs; Noise Canceling Headphones
MeSH Terms: conditions — Delirium; Sleep Deprivation; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Usual Care (No Intervention): Usual Care between 10pm-6am
- Earplugs (Active Comparator): Application of foam earplugs from 10pm-6am nightly for seven nights or until ICU discharge.
  Interventions: Device: Foam Earplugs
- Earplugs and Headphones (Active Comparator): Foam Earplugs and Noise canceling headphones applied from 10pm-6am nightly for 7 nights or until ICU discharge.
  Interventions: Device: Foam Earplugs; Device: Noise Canceling Headphones

INTERVENTIONS:
Device: Foam Earplugs — Standard Foam Earplugs applied from 10pm-6am nightly. (Sperian Technologies, manufacturer)
  Arms: Earplugs; Earplugs and Headphones
Device: Noise Canceling Headphones — Noise Canceling headphones applied over the ears between 10pm-6am nightly. Model is Bose QuietComfort 15, manufactured by Bose Technologies.
  Arms: Earplugs and Headphones

SUMMARY:
This study seeks to examine the effects of overnight noise reduction in critically ill patients who are receiving mechanical ventilation. The investigators will randomly place subjects into one of three groups: 1) usual care 2) overnight earplugs 3) overnight earplugs and noise-canceling headphones. The investigators will monitor for safety, and will measure the amount of delirium experienced by subjects, record the amount of sedating and painkilling medicines required, and measure sleep quality during the study, among other information. The investigators will also measure noise levels experienced by patients in each group. The investigators predict that the use of overnight noise reduction will be safe and will reduce the amount of delirium by improving the quality of sleep in critically ill patients.

DETAILED DESCRIPTION:
Delirium is an acute confusional state defined by fluctuating mental status, inattention, and either disorganized thinking or an altered level of consciousness. Acute delirium is an increasingly recognized problem in intensive care units (ICUs) in the US and worldwide. ICU Delirium has been estimated to occur in as many as 50 to 80 percent of ICU patients. Delirium in the ICU has been associated with worsened clinical outcomes such as prolonged hospitalization and death [1-4]. Although noise has been shown to negatively influence sleep in the ICU, and sleep disturbance is a recognized contributor to ICU delirium[1-2, 4], there is no well-established link between ICU noise levels and the development of ICU delirium. Optimal strategies for the prevention and treatment of ICU delirium are yet to be defined, and this study will focus on a novel noise-reduction approach which has potential to impact both prevention and treatment [5-8]. Findings will be generalizable to other tertiary care medical intensive care units caring for adult patients.

Objectives Our multidisciplinary team will evaluate the safety and feasibility of direct noise reduction in the Wake Forest University Baptist Medical Center (WFUBMC) Medical Intensive Care Unit (MICU), and any effect on the incidence of ICU delirium.

Methods and Measures Design

* Forty-five (45) patients receiving mechanical ventilation will be randomized to receive either passive direct noise reduction (earplugs), both passive and active direct noise reduction (earplugs and noise-canceling headphones), or no direct noise reduction (usual practice).
* Ambient noise levels and the reduction in noise accomplished by direct noise reduction will be measured according to standardized audiometric techniques.
* Sleep structure, including amount of recovery sleep, will be measured over one night according to standardized polysomnographic (sleep study) techniques
* The incidence of delirium will be assessed as well as multiple other endpoints including but not limited to amount of psychoactive medication prescribed and amount of physical restraints required.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who are admitted to our MICU for at least 24 hours with at least 72 hours' additional expected stay in ICU, and who are mechanically ventilated

Exclusion Criteria:

* severe to profound hearing loss
* baseline use of hearing aids
* eardrum perforation
* severe cerumen impaction
* head or oromaxillofacial trauma
* external ventricular drain or intracranial pressure monitoring devices
* comatose patients who are deemed by their attending physician as unlikely to awaken within 72 hours
* patient status as comfort-measures only
* any other contraindication to the use of earplugs or headphones

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-05; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew C Miles, MD, Study Director — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
de-identified data was shared with another investigator as part of a review and meta-analysis

RESULTS

PARTICIPANT FLOW:
Groups:
- Earplugs: Application of earplugs from 10pm-6am nightly for seven nights or until ICU discharge.
  Foam Earplugs: Standard Foam Earplugs applied from 10pm-6am nightly. (Sperian Technologies, manufacturer)
- Earplugs and Headphones: Earplugs and Noise-canceling headphones applied from 10pm-6am nightly for 7 nights or until ICU discharge.
  Foam Earplugs: Standard Foam Earplugs applied from 10pm-6am nightly. (Sperian Technologies, manufacturer)
  Noise Canceling Headphones: Noise Canceling headphones applied over the ears between 10pm-6am nightly. Model is Bose QuietComfort 15, manufactured by Bose Technologies.
Period: Overall Study
Arm/Group | Usual Care | Earplugs | Earplugs and Headphones
Started | 2 | 3 | 3
Completed | 2 | 3 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Earplugs | Earplugs and Headphones | Total
Number analyzed (Participants) | 2 | 3 | 3 | 8
Age, Continuous [Mean (Full Range); unit: years] | 72 [71 to 73] | 66 [53 to 71] | 56 [40 to 77] | 63 [40 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 2 | 5
  Male | 2 | 0 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 3 | 8
Mean SAPS II [Mean (Full Range); unit: units on a scale] — Severe Acute Physiology Scale II. The SAPS II score is made of 12 physiological variables and 3 disease-related variables. The worst physiological variables were collected within the first 24 hours of ICU admission. The "worst" measurement was defined as the measure that correlated to the highest number of points. The study did not continually calculate SAPS II scores beyond the first 24 hours of ICU admission. The SAPS II score ranges from 0 to 163 points.
  units on a scale | 57.5 [27 to 88] | 40 [22 to 68] | 57.6 [43 to 74] | 51 [22 to 88]

OUTCOME MEASURES:

1. Primary Outcome: Days Free of Delirium or Coma
Time Frame: During the Study Period (Study Days 0-7 while patients were in ICU)
Measure: Mean (Full Range); unit: days
Arm/Group | Usual Care | Earplugs | Earplugs and Headphones
Number analyzed (Participants) | 2 | 3 | 3
days | 0.5 [0 to 1] | 2.3 [0 to 6] | 2 [0 to 4]

2. Secondary Outcome: Noise Attenuation
Description: The reduction in noise experienced by the subject when using the study intervention.
Time Frame: Overnight (10pm-6am) on study day 2 or 3.
Population: Devices were unable to measure noise above 85 dB(A) from the in-ear location; no noise data was collected.
Arm/Group | Usual Care | Earplugs | Earplugs and Headphones
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Sleep Efficiency and Architecture
Description: Staging of sleep with efficiency determined as a ratio of total sleep time/total study time.
Time Frame: Overnight (10pm-6am) on study day 2 or 3
Population: Sleep measurement equipment was not available for use during the study period
Arm/Group | Usual Care | Earplugs | Earplugs and Headphones
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Amount of Sedative Use (Midazolam and Lorazepam)
Time Frame: During the Study Period (Study Days 0-7)
Measure: Mean (Full Range); unit: mg
Arm/Group | Usual Care | Earplugs | Earplugs and Headphones
Number analyzed (Participants) | 2 | 3 | 3
mg
  Midazolam | 5 [0 to 25] | 10.65 [0 to 79.5] | 9.22 [0 to 63.5]
  Lorazepam | 0.21 [0 to 6] | 0.40 [0 to 6.5] | 0.39 [0 to 2]

5. Secondary Outcome: Amount of Analgesic Use
Description: Mean of analgesic daily use
Time Frame: During the Study Period (Study Days 0-7)
Measure: Mean (Full Range); unit: mg
Arm/Group | Usual Care | Earplugs | Earplugs and Headphones
Number analyzed (Participants) | 2 | 3 | 3
mg
  Fentanyl | 0.29 [0 to 0.55] | 0.37 [0 to 2.425] | 0.32 [0 to 2.575]
  Morphine | 0 [0 to 0] | 0 [0 to 0] | 0.03 [0 to 1.5]
  Dilaudid | 0 [0 to 0] | 0 [0 to 0] | 0.07 [0 to 4]
  Hydrocodone | 0 [0 to 0] | 0 [0 to 0] | 0.18 [0 to 5]

6. Secondary Outcome: Amount of Sedative Use (Propofol and Demedetomidine )
Description: Mean of sedative daily use (Propofol and Demedetomidine )
Time Frame: During the Study Period (Study Days 0-7)
Measure: Mean (Full Range); unit: mcg/kg
Arm/Group | Usual Care | Earplugs | Earplugs and Headphones
Number analyzed (Participants) | 2 | 3 | 3
mcg/kg
  Propofol | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Demedetomidine | 1.36 [0 to 13.6] | 0.98 [0 to 9.9] | 0 [0 to 0]

ADVERSE EVENTS:
Arm/Group | Usual Care | Earplugs | Earplugs and Headphones
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes